CLINICAL TRIAL: NCT06413602
Title: Exploring the Synergistic Effects of AIH and FES in Persons With MS
Brief Title: The Synergistic Effects of AIH and FES in Persons With MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Milap Sandhu, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU00221027
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive
Keywords: multiple sclerosis; plasticity; electrical stimulation; NMES; modalities; neuroplasticity; motoneuron; aih; hypoxia; acute intermittent hypoxia
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Hypoxia | interventions — Insemination, Artificial, Homologous

STUDY DESIGN:
Intervention Model Description: randomized, blinded, cross-over study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AIH alone (Experimental): Participants will undergo 30 minutes of AIH.
  Interventions: Other: Acute Intermittent Hypoxia
- NMES alone (Experimental): Participants will undergo repetitive common peroneal nerve stimulation for up to 30 minutes.
  Interventions: Other: Neuromuscular Electrical Stimulation
- Combined AIH and NMES (Experimental): Participants will undergo 30 minutes of AIH. Immediately following, participants will undergo NMES for up to 30 minutes.
  Interventions: Other: Acute Intermittent Hypoxia; Other: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — During AIH, the participant will be equipped with a non-rebreathing face mask, and provided with the AIH intervention. The AIH intervention involves alternating breathing cycles. One cycle involves breathing air with lower oxygen concentration (9-10% oxygen) for 30 and 90 seconds, followed by breathing normal room air (21% oxygen) for a similar duration. This cycle is repeated 15 times in one session. Blood oxygen and heart rate are monitored throughout.
  Other Names: AIH
  Arms: AIH alone; Combined AIH and NMES
Other: Neuromuscular Electrical Stimulation — During NMES, participants will receive electrical stimulation to the common peroneal nerve. Stimulation will be done with a 50% duty cycle, duration of 0.5-1ms for each pulse and a frequency 25-40 Hz. The stimulus intensity will be adjusted to produce approximately 50% of the maximum M-wave (compound muscle action potential) for each participant.
  Other Names: NMES
  Arms: Combined AIH and NMES; NMES alone

SUMMARY:
The purpose of this study is to examine how neuromuscular electrical stimulation (NMES), may synergistically enhance corticospinal excitability in people with relapsing form multiple sclerosis (MS). This is an important intermediate step to evaluate the potential of AIH + NMES as a plasticity-priming strategy for more efficacious interventions for persons with MS. This study will measure ankle torque generation and amplitude of motor evoked potentials (MEPs) using a repeated measures study design in order to better understand the effects of AIH combined with NMES, as compared to only receiving NMES, and only receiving AIH.

DETAILED DESCRIPTION:
NMES: NMES refers to the application of mild electrical stimulation and is often used as an assistive technology for foot drop in MS and other neurologic conditions. The NMES-induced improvement in motor performance appears to be mediated primarily by an increase in corticomotoneuronal excitability. A single session of NMES applied over a peripheral nerve, has been shown to transiently increase net corticospinal excitability (increased MEP amplitude) in both able-bodied individuals and in people with neurological conditions.

AIH: AIH involves breathing brief bouts of low levels of oxygen. Research has found AIH to be a safe and effective intervention resulting in increased ankle strength in people with MS. While AIH has shown potential in enhancing neuroplasticity in people with spinal cord injury (SCI), it has yet to be studied extensively in MS. Preliminary research in the MS population demonstrates that a single session of AIH enhances motor output, increasing voluntary muscle strength by as much as 15-20% within 60 minutes. Over the past decade, studies have found AIH can rapidly enhance neural plasticity in persons with incomplete SCI. AIH activates the serotonergic pathway, leading to increased activity of serotonin receptors and the synthesis of plasticity-related proteins. This plasticity is manifested by a rapid increase in voluntary muscle strength, emerging within 60-90 minutes.

In this study, the investigators will examine how NMES, which has been shown to affect cortical excitability, and AIH, which has been shown to affect corticospinal plasticity, may synergistically enhance corticospinal excitability in people with relapsing form of MS. Foot drop is a common symptom in the diagnosis of MS where the inability to maintain active dorsiflexion during the swing phase of the gait cycle affects walking efficiency, instability, and falls. Seminal studies show that individuals with MS retain the ability to express plasticity even at higher levels of disease burden. This indicates that strategies targeting neuroplasticity can be used to enhance functional recovery and limit the impact of MS disability. The investigators will conduct a randomized, blinded, placebo-controlled, cross-over study in 20 MS patients with established motor deficits and controlled relapse activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing form of MS
* Expanded Disability Status Scale (EDSS) score of at least 3 and no more than 6.5
* Motor Functional Systems Score (FSS) between 2-4
* Relapse free for at least 1 year
* Age ≥18 years and ≤75 years
* Safe to participate in MRI (as indicated via the SRALab MRI questionnaire)
* No change in Dalfampridine dose at least 2 months prior to enrollment

Exclusion Criteria:

* Uncontrolled hypertension or hypotension (outside 140/90 and 90/60 mmHg)
* History of epilepsy or seizures
* Uncontrolled medical problems affecting the lungs (pulmonary diseases including chronic obstructive pulmonary disease), the heart (cardiovascular diseases) or the musculoskeletal system (orthopedic diseases)
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of stroke
* Metal in head (e.g., surgical clips, shrapnel)
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants
* Surgery to the head
* Any non-MS related neurological diseases
* Illnesses that may have caused brain injury
* Unexplained frequent or severe headaches
* Pregnancy in females
* Implanted devices (e.g., pacemakers, medical pumps, brain stimulators)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Motor Evoked Potentials (MEPs) in Ankle Dorsiflexors | Immediately prior to and within 60 minutes after the intervention.
  The MEPs will be elicited by Transcranial Magnetic Stimulation (TMS), a procedure that uses magnetic fields to stimulate nerve cells in the brain.

SECONDARY OUTCOMES:
Ankle Dorsiflexion Torque | Immediately prior to and within 60 minutes after the intervention.
  Maximal volitional ankle dorsiflexion flexion torque will be measured using a strength testing dynamometer (Biodex System 4).
Ankle Dorsiflexion EMG | Immediately prior to and within 60 minutes after the intervention.
  While measuring ankle dorsiflexion torque, the investigators will also record surface electromyography (EMG) from the tibialis anterior muscle during each contraction. Average peak EMG amplitude will be calculated.
Symbol Digit Modalities Test | Immediately prior to and within 60 minutes after the intervention.
  A neurocognitive test that requires individuals to pair specific numbers with given geometric figures within 90 seconds. Both written and oral format will be administered, and scores will be calculated by totaling the number of correct answers for each section.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not currently have a plan to share IPD.